CLINICAL TRIAL: NCT01976897
Title: Effect of the Physiological Angular Position of the Resting Knee on Pressure at the Heel/Surface Interface
Acronym: FlessCare
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2013/EVFN-01; 2013-A01063-42 (Other: RCB number)
Record Dates: First submitted 2013-10-30; First posted 2013-11-06 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Adult, Hospitalized
Keywords: heel - mattress pressure interface; flexion; knee angular position

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- The study population: Only one group is included. See inclusion/exclusion criteria.
  Intervention: Knee flexion measurement 1
  Intervention: Knee flexion measurement 2
  Intervention: Heel - interface pressure measurements
  Interventions: Other: Knee flexion measurement 1; Other: Knee flexion measurement 2; Other: Heel - interface pressure measurements

INTERVENTIONS:
Other: Knee flexion measurement 1 — The angle of knee flexion during resting, supine position is measured by a first person.
Other: Knee flexion measurement 2 — The angle of knee flexion during resting, supine position is measured by a second person.
Other: Heel - interface pressure measurements — The pressure analysis system used is the X Sensor X3 model (Xsensor Technology Corporation, Calgary, Canada). The sensor mat is made up of transducer cells, each measuring 1.6 cm^2. The digital signal is transmitted to a PC via a USB port at a sampling frequency of 10Hz. Before each measurement, the sensor mat is calibrated from 10 to 220 mm Hg, according to the manufacturer's recommendations.
  The sheet of pressure sensors is disposed on the dedicated bed. The patient is then asked to take his/her usual position in the supine position and a latency of 5 minutes is observed. The recording time pressure is then performed for 90 seconds in the optical observing time to adapt to changes in media.

SUMMARY:
The main objective of this study is to evaluate the relationship between the angle of knee flexion in a supine position with joint relaxation (DDPD) and the maximum interface pressure at the heel area (PtAl).

DETAILED DESCRIPTION:
The secondary objectives of this study are:

A. To evaluate the relationship between the angle of flexion of the knee in DDPD and the average pressure throughout the heel area (Pmean).

B. To evaluate the relationship between the angle of flexion of the knee in DDPD and the contact surface of the heel area (Stal) where the pressure is greater than 60 mm Hg.

C. To evaluate the inter-operator concordance for the knee flexion angle measurement in DDPD via photos.

D. To evaluate the inter-operator concordance for skin marks used to measure knee flexion angles in DDPD via photos (only one knee for 30 patients).

E. To evaluate the inta-operator concordance (measures on 2 consecutive days) for skin marks used to measure knee flexion angles in DDPD via photos (for 30 patients).

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is in a stable medical state (no complications within the past 10 days)

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient has had medical complications within the ten days preceding study inclusion
* The patient has a bed-sore or bandages on his/her heels
* The patient has had a lower-limb amputation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of consecutive patients admitted in the functional rehabilitation unit of the Nîmes University Hospital.
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2014-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Measurement 1: Measurement of the knee joint angle (degrees °) in a physiological relaxed position (supine)(via photos of first skin marks). | Day 0
Measurement 2: Measurement of the knee joint angle (degrees °) in a physiological relaxed position (supine)(via photos of first skin marks) | Day 0
Maximum pressure on the heel area (Ptal) | Day 0

SECONDARY OUTCOMES:
Mean pressure over the entire heel area (P mean) | Day 0
Measurement of the contact surface of the heel zone (Stal) having a pressure greater than 60 mmHg | Day 0
Concordance for measurements 1 & 2 for knee flexion angle in a relaxed supine position (via photos) | Day 0
Concordance for skin marks for knee flexion angles between 2 operators for 30 knees. | Day 0
  relaxed, decubitus dorsal position
Intra-operator concordance for skin marks used for measuring knee flexion angle for 30 knees | Day 1
  Relaxed decubitus dorsal position

OTHER OUTCOMES:
Age | Day 0
Sex | Day 0
Weight (kg) | Day 0
Height (cm) | Day 0
Braden risk scale | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Viollet, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France